CLINICAL TRIAL: NCT04416503
Title: Effect of Reflexology on Ankle Brachial Index, Diabetic Peripheral Neuropathy, and Glycemic Control in Elderly Diabetic Individuals
Brief Title: Effect of Reflexology on Diabetic Foot and Glycemic Control in Elderly Diabetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-HSF-SCC-01
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Reflexology; Type 2 Diabetes; Older People
Keywords: Aged; Ankle brachial index; Diabetic neuropathies; Glycated hemoglobin A; Musculoskeletal manipulations
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Foot reflexology was performed for 12 week in the intervention group, whereas the control group continued their routine treatment and follow-up.
  Interventions: Other: Foot reflexology
- Control group (No Intervention): Usual follow-up was done to the control group.

INTERVENTIONS:
Other: Foot reflexology — Foot reflexology was performed for 12 week in the study group,whereas the control group continued their routine treatment and follow-up.
  Arms: Intervention group

SUMMARY:
Background: Glycemic control can be difficult in the elderly with diabetes.Diabetic foot problems characterized by vascular and neuropathy are serious complications. The effectiveness of reflexology has been demonstrated to achieve glycemic control and manage diabetic foot problems.

Objectives: To determine the effect of foot reflexology on ankle brachial index (ABI), diabetic peripheral neuropathy (DPN) and glycemic control in elderly diabetic individuals.

Design: A randomized clinical trial. Settings: An outpatient elderly health center in Turkey. Participants: 48 individuals aged 65 and over enrolled in the elderly health center were included.

Methods: The elderly were randomized into two groups (study, n=24; control,n=24). Foot reflexology was performed for 12 week in the study group, whereas the control group continued their routine treatment and follow-up. Both groups underwent a comprehensive foot examination for evaluating ABI and DPN at baseline and after 12 weeks; furthermore, glycemic control (glycated hemoglobin-HbA1c) was evaluated. An independent two-sample t-test was performed for pre- and post-test between-group comparisons; an effect size analysis was performed to determine the effect of intervention.

DETAILED DESCRIPTION:
Background: Elderly individuals often refer to the health facility with the complications of diabetes as the first reason. Glycemic control can be quite difficult in elderly diabetic individuals compared to other age groups. Diabetic foot problems, leading to progressive problems from circulatory disorders and nervous loss to organ loss, constitute the most serious complications. Foot reflexology has been shown as a useful practice in the management of glycemic control and foot problems in diabetic individuals. Reflexology has been shown to have a positive effect on glycemic control and the management of diabetic foot problems. There are clinical trials of reflexology in Turkey for use in a variety of diseases or conditions, but there are no studies about diabetes or diabetes complications. Therefore, current research is a first in this regard. In this context, this study has been performed to determine the effect of foot reflexology on ABI, DPN, and glycemic control in elderly diabetic individuals.

Design: A randomized clinical trial. Settings: An outpatient elderly health center in Turkey. Participants: 48 individuals aged 65 and over enrolled in the elderly health center were included.

Measures: At baseline, subjective area was collected by participant information form. Glycemic control was evaluated with HbA1c. DPN and ABI assessment were performed by physical examination of the foot at baseline and three months later.

Methods: The elderly were randomized into two groups (study, n=24; control, n=24). Foot reflexology was performed for 12 week in the study group, whereas the control group continued their routine treatment and follow-up. Both groups underwent a comprehensive foot examination for evaluating ABI and DPN at baseline and after 12 weeks; furthermore, HbA1c was evaluated. An independent two-sample t-test was performed for pre- and post-test between-group comparisons; an effect size analysis was performed to determine the effect of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Older than 65 years with type 2 diabetes
* No fractures or open wounds on both lower limbs
* No single or double sided amputation on the lower limbs.

Exclusion Criteria:

* Uncontrolled high blood pressure
* Acute infection with fever
* Acute surgical conditions
* Receiving dialysis treatment
* Being a verbal communication problem related to Alzheimer's or dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Means of Ankle Brachial Index score | 3-month change
  Vascular assessment test to assess peripheral circulation in the lower limbs. The measurement, obtained by dividing the highest ankle arterial pressure (posterior tibial or dorsalis pedis) on the same side by brachial pressure, was evaluated using a 5-10-MHz handheld Doppler device and a blood pressure cuff.
Means of Diabetic peripheral neuropathy score | 3-month change
  Measurement parameter testing whether there is nerve damage due to diabetes by physical examination of the foot. The examination was determined using symptom and disability scores. Symptom scores included questions related to complaints experienced by patients, the location of the complaints, the presence of night or day symptoms, and how the symptoms relieved/subsided. Disability scores were determined with four parameters: vibration sensation (128 Hz tuning fork), pinprick sensation, achilles reflex and sensitivity to touch (Semmes-Weinstein nylon monofilaments 10 g).Participant responses and examination findings were scored according to a guideline and a neuropathy score was obtained for each participant.
HbA1c levels (%) | 3-month change
  Blood test to evaluate glycemic control. Blood sample was collected in EDTA-coated tubes (2 mL of whole) from the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman ÖZSARI, PhD, DR, Study Director — Bolu Provincial Health Directorate
Locations (1):
- Bolu Elderly Health Center, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cicek SC, Demir S, Yilmaz D, Yildiz S. Effect of reflexology on ankle brachial index, diabetic peripheral neuropathy, and glycemic control in older adults with diabetes: A randomized controlled trial. Complement Ther Clin Pract. 2021 Aug;44:101437. doi: 10.1016/j.ctcp.2021.101437. Epub 2021 Jul 4. PMID 34237668